CLINICAL TRIAL: NCT03933215
Title: Cladribine Tablets: Observational Evaluation of Effectiveness and PROs in Suboptimally Controlled Patients Previously Taking Injectable DMDs for RMS (CLICK-MS)
Brief Title: A Study of Suboptimally Controlled Participants Previously Taking Injectable DMDs for RMS (CLICK-MS)
Status: Completed | Type: Observational
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS700568_0078
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cladribine Tablets; Observational; Mavenclad
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cladribine
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — Participants received cladribine tablets as per investigator discretion and as per United States approved label: 3.5 milligram/kilogram (mg/kg) body weight over 2 years, administered as 1 treatment course of 1.75 mg/kg per year.

SUMMARY:
To evaluate the effectiveness, patient-reported outcomes (PROs) and safety of cladribine tablets in participants with relapsing forms of multiple sclerosis (RMS) including relapsing-remitting multiple sclerosis (RRMS) and active secondary progressive multiple sclerosis (aSPMS),who transition to cladribine tablets after suboptimal response to any injectable disease-modifying drugs (DMDs) approved in the United States (US) for RMS in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants greater than or equal to (>=)18 years
* Signed informed consent
* Have diagnosis of RMS including RRMS and aSPMS and satisfy the approved indication for cladribine tablets as per United States Prescribing Information (USPI)
* Have time since diagnosis of RMS of at least 12 months
* Had received their last previous injectable disease-modifying drug (DMD) for at least 3 months
* Have decided to initiate treatment with cladribine tablets during routine clinical care
* Meet criteria as per the approved USPI
* Have access to a valid e-mail address
* In the opinion of the Investigator, experienced suboptimal response (lack of effectiveness, intolerability, poor adherence) to injectable DMD treatment

Exclusion Criteria:

* Have been previously treated with cladribine in any dosing form
* Transitioning from previous injectable DMD solely for administrative reasons such as relocation
* Have comorbid conditions that preclude participation
* Have any clinical condition or medical history noted as contraindication on USPI
* Are currently participating in an interventional clinical trial
* Pregnant or breastfeeding women, women who plan to become pregnant or men whose partner plans to become pregnant during the cladribine treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Multiple Sclerosis and experienced suboptimal response (lack of effectiveness, intolerability, poor adherence) to prior treatment with an injectable DMD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., the biopharmaceutical division of Merck KGaA, Darmstadt, Germany
Locations (18):
- United States (18):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - HCA Research Institute, Englewood, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Prairie Education & Research, Springfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - College Park Family Care Center, Overland Park, Kansas
  - The Elliot Lewis Center for Multiple Sclerosis Care, LLC, Wellesley, Massachusetts
  - UMASS - Neurology, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Minneapolis Clinic of Neurology - Neurology, Minneapolis, Minnesota
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Neurology Center of San Antonio, San Antonio, Texas
  - Blacksburg Neurology, PC, Christiansburg, Virginia
  - Neurological Associates, Richmond, Virginia
  - VCU Medical Center - Pediatric Neurology, Richmond, Virginia
  - Sentara Ambulatory Care Center, Virginia Beach, Virginia
  - MS Center of Evergreen, Kirkland, Washington

REFERENCES:
- [Background] Miravalle AA, Katz J, Robertson D, Hayward B, Harlow DE, Lebson LA, Sloane JA, Bass AD, Fox EJ. CLICK-MS and MASTER-2 Phase IV trial design: cladribine tablets in suboptimally controlled relapsing multiple sclerosis. Neurodegener Dis Manag. 2021 Apr;11(2):99-111. doi: 10.2217/nmt-2020-0059. Epub 2021 Feb 1. PMID 33517769
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0078
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cladribine
Started | 100
Treated | 62
Completed | 34
Not Completed | 66
Not completed — Other | 6
Not completed — Sponsor decision | 5
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 6
Not completed — Enrolled but not treated | 38

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Arm/Group | Cladribine
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 52
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).
Time Frame: Baseline (Month 0) up to 24 Months
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of cladribine tablets. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 51
relapses per year | 0.02 [0.000 to 0.059]

2. Secondary Outcome: Change From Baseline in 14-Item Treatment Satisfaction Questionnaire for Medication (TSQM-14) Score at Month 6, 12 and 24
Description: The TSQM-14 was a participant-rated scale used to assess subjective satisfaction with medication. The TSQM has 14 questions that assesses participants' global satisfaction level with their treatment in 4 domains: side effects (There are 5 questions in the side effects domain, however one of them is a Yes/No question and there are 4 sub-components, hence a maximum score of 20), effectiveness (3 questions), global satisfaction (3 questions), and convenience (3 questions). All questions are scored from 1 (least satisfied) to 5 or 7 (most satisfied). The total score is summed for each domain to obtain: side effects (1-20), effectiveness (1-21), global satisfaction (1-17), and convenience (1-21), using transformed scores between 0 and 100. Lower total scores in each domain indicate dissatisfaction with the study medication and higher total scores indicate satisfaction.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of cladribine tablets. Here, "overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at each specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 10
units on a scale
  Global Satisfaction: change at Month 6 | 32.9 (29.01)
  Global Satisfaction: change at Month 12: number analyzed (Participants) | 9
  Global Satisfaction: change at Month 12 | 26.2 (21.43)
  Global Satisfaction: change at Month 24: number analyzed (Participants) | 1
  Global Satisfaction: change at Month 24 | 7.1 (NA) — The standard deviation could not be calculated with data from only 1 participant.
  Effectiveness: change at Month 6 | 24.4 (23.45)
  Effectiveness: change at Month 12: number analyzed (Participants) | 9
  Effectiveness: change at Month 12 | 7.4 (35.13)
  Effectiveness: change at Month 24: number analyzed (Participants) | 1
  Effectiveness: change at Month 24 | -5.6 (NA) — The standard deviation could not be calculated with data from only 1 participant.
  Side Effects: change at Month 6 | -8.8 (41.37)
  Side Effects: change at Month 12: number analyzed (Participants) | 9
  Side Effects: change at Month 12 | -18.1 (24.69)
  Side Effects: change at Month 24: number analyzed (Participants) | 1
  Side Effects: change at Month 24 | 0.0 (NA) — The standard deviation could not be calculated with data from only 1 participant.
  Convenience: change at Month 6 | 35.0 (21.44)
  Convenience: change at Month 12: number analyzed (Participants) | 9
  Convenience: change at Month 12 | 24.7 (19.66)
  Convenience: change at Month 24: number analyzed (Participants) | 1
  Convenience: change at Month 24 | 33.3 (NA) — The standard deviation could not be calculated with data from only 1 participant.

3. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Score at Month 6, 12 and 24
Description: SF-36 was a multipurpose, participant completed, short-form health survey with 36 questions that consists of an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. Physical component summary (PCS) is mostly contributed by physical function (PF), role physical (RP), bodily pain (BP), and general health (GH). Mental component summary (MCS) is mostly contributed by mental health (MH), role emotional (RE), social function (SF), and vitality (VT). Each component on the SF-36 item health survey is scored from 0 (best) to 100 (worst). Total score ranges from 0-100 for each component summary (i.e., PCS and MCS), where higher scores are associated with less disability and better quality of life.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 15
units on a scale
  PCS: Change at Month 6: number analyzed (Participants) | 13
  PCS: Change at Month 6 | 4.1 (6.90)
  PCS: Change at Month 12 | -0.4 (5.68)
  PCS: Change at Month 24: number analyzed (Participants) | 1
  PCS: Change at Month 24 | 1.9 (NA) — The standard deviation could not be calculated with data from only 1 participant.
  MCS: Change at Month 6: number analyzed (Participants) | 13
  MCS: Change at Month 6 | 0.9 (7.66)
  MCS: Change at Month 12 | 0.3 (8.05)
  MCS: Change at Month 24: number analyzed (Participants) | 1
  MCS: Change at Month 24 | -2.5 (NA) — The standard deviation could not be calculated with data from only 1 participant.

4. Secondary Outcome: Change From Baseline in Modified Fatigue Impact Scale - 5-item Version (MFIS-5) Total Score at Month 6, 12 and 24
Description: MFIS-5 is a modified form of the Fatigue Impact Scale that consists of 5 questions that assess the impact of fatigue on physical, cognitive, and psychosocial functioning, with 5 response levels ranging from 0 to 4, where 0 = (Never), 1 = (Rarely), 2 = (Sometimes), 3 = (Often), 4 = (Almost always). Total scores range from 0 to 20, with higher scores representing a greater impact of fatigue.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 14
units on a scale
  Change at Month 6: number analyzed (Participants) | 12
  Change at Month 6 | -2.1 (3.42)
  Change at Month 12 | 0.4 (4.73)
  Change at Month 24: number analyzed (Participants) | 1
  Change at Month 24 | 0.0 (NA) — The standard deviation could not be calculated with data from only 1 participant.

5. Secondary Outcome: Change From Baseline in 7-Item Beck-Depression Inventory-Fast Screen (BDI-FS) Total Score at Month 6, 12 and 24
Description: The 7 items BDI-FS is a self-report inventory for measuring the severity of depression on a 7-item scale. The BDI-Fast Screen is scored by summing all of the highest ratings for each of the 7 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 21. Higher scores indicate greater symptom severity.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 13
units on a scale
  Change at Month 6 | -1.3 (3.09)
  Change at Month 12 | -0.1 (3.04)
  Change at Month 24: number analyzed (Participants) | 2
  Change at Month 24 | -1.0 (2.83)

6. Secondary Outcome: Change From Baseline in Percent Work Time Missed Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-items validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percent work time missed (absenteeism) was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Cladribine
Number analyzed (Participants) | 13
percentage of work time missed
  Change at Month 6 | 3.1 (16.37)
  Change at Month 12 | -6.3 (28.64)
  Change at Month 24: number analyzed (Participants) | 2
  Change at Month 24 | 0.0 (0.00)

7. Secondary Outcome: Change From Baseline in Percent Impairment While Working Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-items validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percentage of impairment while working (presentisms) was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Cladribine
Number analyzed (Participants) | 13
percentage of impairment while working
  Change at Month 6: number analyzed (Participants) | 7
  Change at Month 6 | -11.4 (6.90)
  Change at Month 12: number analyzed (Participants) | 10
  Change at Month 12 | -5.0 (22.24)
  Change at Month 24: number analyzed (Participants) | 1
  Change at Month 24 | 0.0 (NA) — The standard deviation could not be calculated with data from only 1 participant.

8. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-items validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in total percentage of work impairment (absenteeism and presentisms) were reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Cladribine
Number analyzed (Participants) | 13
percentage of overall work impairment
  Change at Month 6: number analyzed (Participants) | 7
  Change at Month 6 | -5.1 (18.73)
  Change at Month 12: number analyzed (Participants) | 10
  Change at Month 12 | -6.1 (19.99)
  Change at Month 24: number analyzed (Participants) | 1
  Change at Month 24 | 0.0 (NA) — The standard deviation could not be calculated with data from only 1 participant.

9. Secondary Outcome: Change From Baseline in Percent Activity Impairment Assessed by 6-Item Work Productivity Activity Impairment- Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-items validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percent activity impairment was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Cladribine
Number analyzed (Participants) | 13
percentage of activity impairment
  Change at Month 6 | -10.0 (10.00)
  Change at Month 12 | -7.7 (21.27)
  Change at Month 24: number analyzed (Participants) | 2
  Change at Month 24 | -5.0 (7.07)

10. Secondary Outcome: Change From Baseline in Patient Determined Disease Steps (PDDS) Scale Total Score at Month 6, 12 and 24
Description: PDDS scale developed to assess the disability in Multiple Sclerosis (MS) participants and in assessing disease progression that focuses mainly on how participants walk. PDDS scale ranges from 0 to 8, where 0 = normal; 1 = mild disability; 2 = moderate disability; 3 = gait disability; 4 = early cane; 5 = late cane; 6 = bilateral support; 7 = wheelchair/scooter and 8 = bedridden. A higher score represented higher level of disability.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of cladribine tablets. Here, "overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 26
units on a scale
  Change at Month 6 | -0.2 (0.69)
  Change at Month 12: number analyzed (Participants) | 22
  Change at Month 12 | -0.3 (0.72)
  Change at Month 24: number analyzed (Participants) | 14
  Change at Month 24 | -0.1 (1.17)

11. Secondary Outcome: Number of Participants With Adherence to Cladribine as Assessed by Modified Versions of the Multiple Sclerosis Treatment Adherence Questionnaire (MS-TAQ)
Description: 7 Treatment adherence questions, based on MS-TAQ, were developed to determine level of adherence as well as identify barriers to adherence for MS participants taking DMDs. 1.What treatment week of cladribine (Clad.) tablets (tab.) did you most recently complete? 2.How many Clad. tab. were you supposed to take during this treatment week? 3.Did you miss/forget to take any Clad. tab. during this treatment week? 4. How many Clad. tab. did you miss/ forget to take? 5.How important were following factors in missing/forgetting to take a dose? (scale from 0-3, where, 0=Not important at all and 3=Extremely important). 6.Overall, how hard/easy do you feel it is to take Clad. tab. as recommended by your physician during your treatment week? (scale from 1- 5, where 1=Extremely easy and 5=Extremely hard). 7.How satisfied are you with how things have been with your Clad. tab. treatment during your treatment week? (scale from 1-5, where 1=Not satisfied at all and 5=Completely satisfied).
Time Frame: Baseline (Month 0) and Months 1, 2, 13 and 14
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of cladribine tablets. Here, "overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. "Number of participants analyzed at timepoint" signifies those participants who were evaluable for this outcome measure at each specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 40
Participants
  At Baseline | 28
  Month 1: number analyzed (Participants) | 38
  Month 1 | 38
  Month 2: number analyzed (Participants) | 38
  Month 2 | 38
  Month 13: number analyzed (Participants) | 22
  Month 13 | 21
  Month 14: number analyzed (Participants) | 18
  Month 14 | 18

12. Secondary Outcome: Percentage of Participants Who Experienced Relapse at Months 12 and 24
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days). Percentage of participants who experienced relapse at Months 12 and 24 were reported.
Time Frame: Months 12 and 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 62
percentage of participants
  Month 12 | 1.6
  Month 24 | 1.6

13. Secondary Outcome: Annualized Relapse Rate (ARR) at Month 12
Description: as for outcome 1
Time Frame: At Month 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 51
relapses per year | 0.01955 [0.0 to 0.1]

14. Secondary Outcome: Percentage of Participants Who Experienced Relapse Associated With Hospitalization
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days). Percentage of participants who experienced relapse associated with hospitalization at Months 12 and 24 were reported.
Time Frame: Months 12 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 51
percentage of participants
  Month 12 | 0.0
  Month 24 | 0.0

15. Secondary Outcome: Annualized Relapse Rate (ARR) Associated With Hospitalization at Months 12 and 24
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days). ARR associated with hospitalization at Months 12 and 24 were reported.
Time Frame: Months 12 and 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 51
relapses per year
  Month 12 | 0.0 [0.0 to NA] — The upper limit of 95% confidence interval was not calculated as none of the participant had relapse.
  Month 24 | 0.0 [0.0 to NA] — The upper limit of 95% confidence interval was not calculated as none of the participant had relapse.

16. Secondary Outcome: Percentage of Participants Who Experienced Relapse Associated With Glucocorticoid Use
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).Percentage of participants who experienced relapse associated with glucocorticoid use at Months 12 and 24 were reported.
Time Frame: Months 12 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 51
percentage of participants
  Month 12 | 0.0
  Month 24 | 0.0

17. Secondary Outcome: Annualized Relapse Rate (ARR) Associated With Glucocorticoid Use at Months 12 and 24
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days). ARR associated with glucocorticoid use at Months 12 and 24 were reported.
Time Frame: Months 12 and 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 51
relapses per year
  Month 12 | 0.0 [0.0 to NA] — The upper limit of 95% confidence interval was not calculated as none of the participant had relapse.
  Month 24 | 0.0 [0.0 to NA] — The upper limit of 95% confidence interval was not calculated as none of the participant had relapse.

18. Secondary Outcome: Number of Previous Disease-Modifying Drugs (DMD) Received for Multiple Sclerosis (MS) at Baseline
Description: Number of previous DMD received by participants with MS were reported.
Time Frame: At Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: number of DMDs received
Arm/Group | Cladribine
Number analyzed (Participants) | 62
number of DMDs received | 1.9 (1.14)

19. Secondary Outcome: Number of Participants Who Received At Least One Concomitant Medication
Description: Number of participants who received at least one concomitant medication were reported.
Time Frame: Baseline up to Month 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 62
Participants | 60

20. Secondary Outcome: Percentage of Participants Who Discontinued Cladribine Tablets
Description: Percentage of participants who discontinued cladribine tablets were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 62
percentage of participants | 32.3

21. Secondary Outcome: Elapsed Time to Discontinuation After First Dose of Cladribine Tablets
Description: Elapsed time to discontinuation after first dose of cladribine tablets was reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 62
months | 13.2 [12.2 to 14.1]

22. Secondary Outcome: Number of Doses Received by Participants as Per United States Prescribing Information
Description: Number of doses received by participants as per United States prescribing information were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: number of doses received
Arm/Group | Cladribine
Number analyzed (Participants) | 62
number of doses received | 28.00 [18.00 to 34.00]

23. Secondary Outcome: Percentage of Participants With Treatment Compliance as Per United States Prescribing Information
Description: Treatment compliance was defined as total actual number of cladribine tablets / total planned number of cladribine tablets.
Time Frame: Baseline (Month 0) up to 24 Months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 62
percentage of participants | 82.3

24. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs) and Adverse Events of Special Interest (AESIs)
Description: A serious adverse event (SAE) is an adverse event (AE) that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or is otherwise considered medically important. An ADR is a response to a medicinal product which is noxious and unintended. An AESI is an AE of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor can be appropriate.
Time Frame: Baseline (Month 0) up to 24 months
Population: The Safety Analysis Set (SAF) included all participant enrolled in the study who have received at least 1 dose of cladribine tablets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 62
Participants
  SAE | 3
  ADR | 18
  AESI | 9

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months
Arm/Group | Cladribine
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 3/62
Other Adverse Events (participants affected / at risk) | 34/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine (N=62)
Gastritis (Gastrointestinal disorders) | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Low absolute lymphocyte count (Investigations) | 1
Suspected infection of the kidney (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine (N=62)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 9
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Thyroid disorder (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 5
Croup infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Foot fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 1
Oedema peripheral (General disorders) | 1
Bacterial vulvovaginitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Borderline personality disorder (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
There are methods to adjustment for missing-not-at-random, but these methods are varied and inconsistent, especially with high missingness. Knowing we have low counts for many outcomes, we reported the data that we have, accepting that there will be patients with missing data who are missing assessments due to sickness or other non-random reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must be notified of plans to present or publish data. Presentations and/or publications require pre-submission review and approval by sponsor. Sponsor maintains right to delay publication to protect IP rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03933215/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03933215/SAP_001.pdf